CLINICAL TRIAL: NCT05608122
Title: Establishment of Online Registration Platform for Unruptured Intracranial Aneurysms Based on Regional Medical Centers in China and Population Follow-up Study (Phase Ⅱ)
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Wang Shuo, Department of neurosurgery, Beijing Tiantan Hospital
Other Study IDs: KY-2021-110-01
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-11

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysm; Artificial Intelligence
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- unstable intracranial aneurysms: Unstable intracranial aneurysms are defined as the intracranial aneurysms that grows or ruptures.
  Interventions: Other: Obervation
- stable intracranial aneurysms: Stable intracranial aneurysms are defined as the intracranial aneurysms that have no significant morphological changes.
  Interventions: Other: Obervation

INTERVENTIONS:
Other: Obervation — This study is an observational study without any intervention
  Groups: unstable intracranial aneurysms
Other: Obervation — This study is an observational study without any intervention
  Groups: stable intracranial aneurysms

SUMMARY:
Intracranial aneurysm is the main cause of subarachnoid hemorrhage, and the incidence of subarachnoid hemorrhage in Chinese population is about 5%. The intervention of unruptured intracranial aneurysms is controversial because of its great harm after natural rupture and bleeding, and about a quarter of patients still have poor prognosis through existing invasive treatment methods. How to accurately determine the instability risk of unruptured intracranial aneurysms is the key to resolve this controversy.

In previous studies, the stability of intracranial aneurysms involves many characteristics, and the sample size is small. Most of them are retrospective studies and studies on the status after change (rupture/growth). Therefore, the relevant risk factors are not clear at present, and there is still a lack of reliable prediction model. Based on the above facts, this study proposed based on the national hundred regional medical institutions set up the network registration platform of unruptured intracranial aneurysms, real time and openness of Internet, through the way of case resource sharing build unruptured intracranial aneurysm queue, collecting clinical characteristics, imaging features, hemodynamic detection of biological samples and the results of the analysis data, And observe them for two years. The artificial intelligence platform of Tonglian Medical Health was used to integrate and analyze and learn all the data, and then the risk factors related to the stability of intracranial aneurysms within two years were obtained, and the stability prediction model of unruptured intracranial aneurysms was constructed. This study will build the largest network registration platform and population follow-up cohort of unruptured intracranial aneurysms in China, and put forward a prediction model for the stability of unruptured intracranial aneurysms by integrating the multi-dimensional factors of intracranial aneurysms, so as to provide a powerful auxiliary judgment tool for the clinical decision-making of this disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. At least one unruptured intracranial aneurysm was found by CTA;
3. No relevant symptoms, receiving non-operative and conservative observation treatment;
4. Signing the informed consent.

Exclusion Criteria:

1. Other cerebrovascular structural lesions (such as cerebrovascular malformation and arteriovenous fistula) or craniocerebral tumors;
2. Fusiform or dissecting aneurysms;
3. Traumatic, mycotic and atrial myxoma associated aneurysms;
4. Suffering from systemic connective tissue diseases, such as polycystic kidney disease;
5. Expectant survival of no more than 3 years due to other diseases or poor general conditions;
6. Patients refuse to follow up or cannot communicate with them due to mental diseases;
7. Pregnant women or participating in other aneurysm related studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 3740 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Aneurysm rupture | 2 years

SECONDARY OUTCOMES:
Aneurysm growth | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes